CLINICAL TRIAL: NCT00862290
Title: Diagnostic and Predictive Value of Circulating microRNAs During Sepsis
Brief Title: Circulating microRNAs as Biomarkers of Sepsis
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, M.D., Changhai Hospital
Other Study IDs: microRNA_sepsis
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Sepsis
Keywords: sepsis; microRNA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood of septic patients is collected on the second day when they are diagnosed with sepsis in ICU. Blood of SIRS patients is collected on the second day when they are diagnozed with SIRS after cardiac surgery with cardiopulmonary bypass.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- sepsis group: Patients who develop sepsis in the ICU
- SIRS group: Patients who develop SIRS after cardiac surgery with cardiopulmonary bypass
- control group: normal healthy volunteers

SUMMARY:
MicroRNA has been demonstrated to play a crucial role in regulating cell processes. Recently, microRNA was identified to exist in human serum or plasma, and it might be related to certain diseases. Several microRNAs are involved in sepsis, such as miR-146, miR-155, and so on. But whether serum miR-146 is present in serum of septic patients remains unknown. The present study was designed to identify the existence of specific microRNAs, which might be new markers for sepsis and its prognosis.

ELIGIBILITY:
Inclusion Criteria:

* patients who develop sepsis and undergo abdominal surgery
* patients who develop SIRS after cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* patients with a primary diagnosis of acute pancreatitis
* patients with cirrhosis or renal dysfunction
* patients with dyscrasia
* patients with autoimmunity diseases
* patients with severe cardiac and pulmonary diseases
* patients with hematological diseases
* patients who had organ dysfunction after cardiac surgery with cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who develop sepsis and SIRS
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Relative amount of circulating microRNAs | On the second day of diagnosis of sepsis in ICU

SECONDARY OUTCOMES:
Serum levels of CRP and IL-6 | On the second day of diagnosing sepsis
Apache II score and death | On the second day of diagnosis of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Ke-ming Zhu, M.D., Principal Investigator — Department of Anesthesiology and Intensive Care Unit
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Result] Wang JF, Yu ML, Yu G, Bian JJ, Deng XM, Wan XJ, Zhu KM. Serum miR-146a and miR-223 as potential new biomarkers for sepsis. Biochem Biophys Res Commun. 2010 Mar 26;394(1):184-8. doi: 10.1016/j.bbrc.2010.02.145. Epub 2010 Feb 24. PMID 20188071